CLINICAL TRIAL: NCT05264233
Title: The Acute Effects of Meals Rich in Saturated or Unsaturated Fatty Acids on Postprandial Lipaemia in Healthy Men
Acronym: CocoHeart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, Director of Hugh Sinclair Unit, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 19/30
Record Dates: First submitted 2021-12-16; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Cardiovascular Risk Factor
Keywords: Coconut oil; Postprandial lipaemia; Platelet function; Gastric emptying; Appetite
MeSH Terms: interventions — Coconut Oil; Butter; Plant Oils

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Meal rich in coconut oil (Active Comparator): Participants will be asked to consume a breakfast (0 minute) and lunch (330 minute) rich in coconut oil
  Interventions: Dietary Supplement: Coconut oil
- Meal rich in butter (Active Comparator): Participants will be asked to consume a breakfast (0 minute) and lunch (330 minute) rich in butter
  Interventions: Dietary Supplement: Butter
- Meal rich in vegetable oil (Active Comparator): Participants will be asked to consume a breakfast (0 minute) and lunch (330 minute) rich in vegetable oil
  Interventions: Dietary Supplement: Vegetable oil

INTERVENTIONS:
Dietary Supplement: Coconut oil — 50 g of coconut oil will be added to the test meal for breakfast and 30 g of coconut oil will be added to the test meal for lunch
  Arms: Meal rich in coconut oil
Dietary Supplement: Butter — 50 g of butter will be added to the test meal for breakfast and 30 g of butter will be added to the test meal for lunch
  Arms: Meal rich in butter
Dietary Supplement: Vegetable oil — 50 g of vegetable oil will be added to the test meal for breakfast and 30 g of vegetable oil will be added to the test meal for lunch
  Arms: Meal rich in vegetable oil

SUMMARY:
Current dietary recommendations suggest that lowering intake of saturated fats or replacing it with unsaturated fats will decrease the risk of developing cardiovascular disease. Coconut oil has gained popularity in recent years but it contains 90% saturated fat, which has higher percentage of saturated fat than butter. To date, only limited studies have determined the acute effects of meals containing coconut oil on blood lipids, but findings are inconsistent. Therefore, further studies are needed to address this knowledge gap and compare the postprandial effects of test meals rich in coconut oil with other sources of saturated fatty acids such as butter and unsaturated fatty acids (vegetable oils). A cross-over, double-blind, randomised acute postprandial study will be conducted in 15 healthy men. Participants will be assigned to consume the test meals rich in saturated or unsaturated fatty acids in random order on 3 separate occasions, with 3-4 weeks between each study visit. Participants will be provided with breakfast (toast with jam and milkshake, 50g fat) and lunch (toast with jam and milkshake, 30g fat). The anthropometric, blood pressure, arterial stiffness, and breath samples will be taken for each study visit. Blood samples will be collected for the measurement of fasting lipids, glucose, insulin, inflammatory markers, whole blood culture as well as blood clotting. Breath samples are collected for the measurement of gastric emptying as well as assessment of satiety using questionnaires (100 mm visual analogue scale) completed throughout the day. The findings from this study will contribute to the evidence base on how consuming meals rich in coconut oil influence the level of blood lipids as well as other biomarkers for cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* Aged between 30 to 70 years
* Serum triacylglycerol < 2.3 mmol/l
* Body mass index between 19-32 kg/m2
* Total cholesterol < 7.5 mmol/l

Exclusion Criteria:

* Females
* Smokers
* Medical history of myocardial infarction or stroke in the past 12 months
* Diabetes (defined as fasting glucose > 7.0 mmol/l) or other endocrine disorders
* Kidney, liver, pancreas or gastrointestinal disorder
* Hypertension (blood pressure > 140/90 mmHg), cancer, medication for hyperlipidaemia (e.g. statins), hypertension or, inflammation
* Anaemia (<130 g/L haemoglobin)
* Taking any dietary supplements known to influence lipids/gut microbiota (e.g. plant stanols, fish oil, phytochemicals, natural laxatives, probiotics and prebiotics)
* Drinking in excess of 14 units of alcohol per week
* Planning on a weight-reducing regime
* Parallel participation in another dietary intervention study
* Any other unusual medical history or diet and lifestyle habits or practices that would preclude volunteers from participating in a dietary intervention and metabolic study

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in postprandial triacylglycerol | Acute study: taken at 0 (baseline), 30, 60, 90, 120, 180, 240, 300, 330, 360, 390, 420, 480 minutes
  Triacylglycerol

SECONDARY OUTCOMES:
Fasting blood lipids | Acute study: taken at 0 (baseline)
  Total cholesterol, high density lipoprotein cholesterol, low density lipoprotein cholesterol
Change from baseline in postprandial non-esterified fatty acids | Acute study: taken at 0 (baseline), 30, 60, 90, 120, 180, 240, 300, 330, 360, 390, 420, 480 minutes
  Non-esterified fatty acids
Change from baseline in postprandial insulin | Acute study: taken at 0 (baseline), 30, 60, 90, 120, 180, 240, 300, 330, 360, 390, 420, 480 minutes
  Insulin
Change from baseline in postprandial vascular stiffness | Acute study: taken at 0 (baseline), 150, 315, 465 minutes
  Measured via pulse wave assessment using the Mobil-O-graph device
Change from baseline in postprandial blood pressure | Acute study: taken at 0 (baseline), 180, 300, 480 minutes
  Systolic and diastolic blood pressure
Change from baseline in postprandial thrombin generation | Acute study: taken at 0 (baseline), 180, 330, 480 minutes
  Thrombin generation
Change from baseline in postprandial gastric emptying | Acute study: taken at 15 minutes intervals between 0 min (baseline) and 480 minutes
  Assessed using gas chromatography-mass spectrometry
Appetite rating | Acute study: taken at 30 minutes intervals after the test meals up to 8 hours
  Assessed using 100 mm visual analogue questionnaire
Change from baseline in postprandial gut hormones | Acute study: taken at 0 (baseline), 30, 60, 120, 240, 330, 360, 390 & 480 minutes
  Ghrelin, peptide YY, gastric inhibitory polypeptide, glucagon-like peptide-1
Change from baseline in postprandial endothelial activation | Acute study: taken at 0 (baseline),180, 300 and 420 minutes
  E-selectin, P-selectin, vascular cell adhesion molecule 1, intercellular adhesion molecule-1
Change from baseline in postprandial cytokine | Acute study: taken at 0 (baseline),180, 300 and 420 minutes
  Interleukin 6, interleukin 1 beta, interleukin 10, tumour necrosis factor alpha, C-C motif chemokine ligand 5, C-X-C motif chemokine ligand 5
Weight | Acute study: taken at 0 (baseline)
  Body mass index will be calculated (kg/ height in m^2)
Body composition | Acute study: taken at 0 (baseline)
  Fat mass, fat free mass, trunk fat, trunk fat mass, trunk fat free mass
Habitual diet assessment | Prior to the start of the study
  4-day food diary

OTHER OUTCOMES:
Genotyping for apolipoprotein E | Acute study: taken at 0 (baseline)
  Single nucleotide polymorphisms related to the metabolism of dietary fats

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Lovegrove, BSc PhD, Principal Investigator — University of Reading
Locations (1):
- Department of Food and Nutritional Sciences, University of Reading, Reading, Berkshire, United Kingdom

REFERENCES:
- [Derived] Wong G, Clegg ME, Ross D, Lovegrove JA, Jackson KG. Sequential Meals Containing Animal and Plant-Based Saturated Fats Have Differential Effects on Postprandial Gut Hormones but No Impact on Satiety Compared with Unsaturated Fats in Generally Healthy Males: Findings from the Randomized Controlled Crossover CocoHeart Study. J Nutr. 2025 Jul 1;155(9):3020-9. doi: 10.1016/j.tjnut.2025.06.027. Online ahead of print. PMID 40609691